CLINICAL TRIAL: NCT05038436
Title: Influence of a Medical Device (Polyglucosamine L112) on Serum Surrogate Markers of Cholesterol Absorption: a Prospective Placebo-controlled, Randomised, Double-blind Cross-over Study
Brief Title: Influence of Polyglucosamine L112 on Serum Surrogate Markers of Cholesterol Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Collaborators: University Hospital, Bonn (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EXT-202001
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-03

CONDITIONS: Cholesterol Lowering
Keywords: obesity; weight reduction; cholesterol reduction
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: prospective, randomised, double blind, placebo controlled, 2 period crossover, monocenter
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial product (verum and placebo) is labelled and packaged by an authorised body according to randomisation, so that there is only specific numbering according to randomisation on the otherwise identical-looking packs. An emergency envelope, located at the study centre, can be used to unblind in an emergency by the principal investigator or investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyglucosamine L112 (Experimental): composed of (beta-1.4 polymer of D-glucosamine and N-acetyl-D-glucosamine)
  Interventions: Device: Polyglucosamine L112
- Placebo (Placebo Comparator): Dicalcium phosphate, cellulose
  Interventions: Device: Polyglucosamine L112

INTERVENTIONS:
Device: Polyglucosamine L112 — Two tablets once daily per os

SUMMARY:
Obesity is widespread and the number of overweight people has tripled from 1975 to 2016. According to the WHO (World Health Organisation), 1.9 billion adults worldwide are overweight, of which 650 million are obese. Thus, obesity is caused by a balance problem between the amount of food consumed and the energy used. The weighting of the diet in favour of a far too high fat intake also has a negative influence on the fat metabolism.

Obesity is associated with a number of secondary diseases, such as diabetes mellitus, increased inflammatory parameters in the blood and a higher risk of heart attack and stroke. These secondary diseases reduce the quality and duration of life of the person affected.

In animal studies, polyglucosamine was found to have a cholesterol-lowering effect. In human studies conducted over 3 and 12 months, formoline L112 was shown to lower LDL levels in the blood.

For research purposes, the present study will focus on investigating whether the intake of polyglucosamine L112 leads to a reduction in cholesterol intake from food, which should result in a reduced fat and thus calorie intake.

DETAILED DESCRIPTION:
In the present study, the influence of polyglucosamine L112 on cholesterol absorption in humans is to be investigated in more detail.

For this purpose, the subjects undergo two randomised study periods in a crossover design: first, there is a 2-week run-in phase, during which baseline values are collected without influence, then the subjects undergo two identical study periods, during which the subjects randomly take either polyglucosamine L112 or placebo twice a day. The study periods are separated by a two-week washout phase. After two weeks, a final examination takes place.

Throughout the course of the study, lipids in the serum are measured regularly. In order to examine cholesterol absorption, however, it is not sufficient to determine the cholesterol levels in the blood, as reduced absorption is physiologically compensated for by increased endogenous synthesis.

In the present study, the plant sterol campesterol, which is absorbed from the intestine like cholesterol, is determined as a surrogate marker for cholesterol absorption. At the same time, a surrogate marker for endogenous cholesterol synthesis is determined with lathosterol, which behaves like the endogenously synthesised cholesterol in terms of concentration. However, campesterol must also be set in relation to cholesterol via the campesterol-cholesterol quotient, since the concentration of campesterol is also dependent on the concentration of LDL lipoproteins as transport molecules, which reacts in the same way as the cholesterol concentration. Accordingly, a lower value of the campesterol-cholesterol quotient indicates reduced cholesterol absorption.

The values corrected for total cholesterol then give an overview of the endogenous cholesterol synthesis for the cholesterol precursors, that of the plant sterols via the cholesterol resorption rate in the small intestine and that of the oxysterols via the bile acid synthesis rate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥ 18 years and ≤ 65 years of age at the time of the screening examination.
* Written documented informed consent and consent to participate in the study.
* Body weight must be ≥ 75 kg at the time of the screening examination.
* Balanced omnivorous diet
* Subjects who are able to follow study instructions and are likely to attend all required study visits (compliance)
* Women of childbearing age must use a reliable method of contraception during treatment
* Negative pregnancy test

Exclusion Criteria:

* BMI < 20 and > 30
* Subject is unable to understand the scope, significance and consequences of this clinical trial
* known hypersensitivity to crustaceans or any of the ingredients of polyglucosamine L112
* concurrent participation in another clinical trial or participation in a clinical trial involving the use of an investigational product for up to 30 days prior to participation in this trial
* known or suspected abuse of medications, drugs, or alcohol
* existing or planned pregnancy or lactation
* not using any contraceptive measure
* previous or active malignant disease
* liver or kidney dysfunction
* history of or clinical evidence of heart failure
* History of lactose intolerance
* Serum laboratory parameters:
* TSH not within normal range
* Creatinine not within normal range
* Bilirubin not within normal range
* Alkaline phosphatase not within normal range
* ALT/AST > 1.5xULN (upper normal limit)
* LDL cholesterol < 130 and >180 mg/dl
* Triglycerides > 200 mg/dl
* HbA1c > 6.5
* Campesterol in serum > 1 mg/dl
* Intake of food supplements (e.g. Becel Proactive)
* Contraindications for weight-reducing therapy
* Pure vegan diet
* Pure meat diet
* Diabetes mellitus type I and II
* Serious gastrointestinal diseases (ulcerative colitis, Crohn's disease, diverticulitis, short bowel syndrome, gastric ulcer, pronounced irritable bowel syndrome, reflux treated with medication, etc.) and after operations in the gastrointestinal tract (except: appendectomy)
* chronic digestive problems (constipation, constipation, etc.)
* Any other disease or medical treatment that, in the opinion of the investigator, could interfere with the assessment of safety, tolerability or efficacy.
* Current medication
* Lipid-lowering drugs such as statins, fibrates, ezitimib or PCSK9 inhibitors
* Interactions with polyglucosamine L112 are expected with the following medications: lipophilic oral medications such as cerebrally active drugs (including antiepileptics), lipophilic hormones (including the contraceptive pill), lipophilic antibiotics, digitalis, fat-soluble vitamins (A, D, E, K), (poly)unsaturated fatty acids.

Exception: Participation in the study is possible if medicinal products for which an interaction is to be expected or cannot be ruled out can be taken at least 4 hours apart from polyglucosamine L112. I.e. since the test product must be taken with the main meals, participation in the study can only take place if it is not necessary to take it with the two main meals.

* taking proton pump inhibitors
* Long-term medication that reduces bowel activity (e.g. opiates)
* Subjects who are dependent on corticosteroids and who cannot be discontinued in time 10 days before the start of the study.
* Taking vitamin K antagonists or other anticoagulants
* Not taking stable medication that can lead to weight gain (e.g. certain neuroleptics, beta-blockers, psychotropic drugs)
* Taking orlistat
* Deliberate weight reduction >10 kg within the last 5 months
* Unintentional weight reduction within the last 5 months > 5 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Influence of polyglucosamine L112 on dietary cholesterol absorption | 10 weeks
  Comparison of the campesterol-cholesterol quotient taking polyglucosamine L112 versus placebo

SECONDARY OUTCOMES:
Influence of polyglucosamine L112 on surrogate markers of cholesterol | 10 weeks
  Comparison of the ratio of sitosterol to cholesterol (cholesterol absorption)
Influence of polyglucosamine L112 on cholesterol synthesis | 10 weeks
  Comparison of the ratio of lathosterol to cholesterol
Influence of polyglucosamine L112 on bile acid synthesis | 10 weeks
  Comparison of the ratio of 7a- and 27-hydroxycholesterol to cholesterol
Influence of polyglucosamine L112 on neutral fecal sterols | 10 weeks
  Comparison of the content of neutral sterols (cholesterol and bacterial degradation products coprostanol and coprostanone)
Fecal primary and secondary bile acids | 10 weeks
  Comparison of the content of bile acids in the stool (cholic acid, deoxycholic acid, chenodeoxycholic acid, lithocholic acid and ursodeoxycholic acid)
Cholesterol measurements | 10 weeks
  Comparison of total cholesterol (C), HDL-C, and LDL-C and triglycerides in serum
Change in body weight | 10 weeks
  Comparison of body weight taking polyglucosamine L112 versus placebo
Safety and tolerability (i.e. incidents of treatment-emergent adverse events) of polyglucosamine L112 | 10 weeks
  Comparison of incidence of adverse events with polyglucosamine L112 versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Martin Coenen, MD, Principal Investigator — University Hospital Bonn, Germany
Locations (1):
- Phase I-Unit, Study Center Bonn (SZB), University Hospital Bonn, Bonn, North-Rhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No